CLINICAL TRIAL: NCT05249868
Title: Multicentre Study on the Impact of the SARS-CoV-2 Pandemic on the Health Status of People Aged 75 and Over and Their Caregivers (CUIDAMOS+75 Project)
Brief Title: Impact of the COVID-19 Pandemic on the Health Status of People Aged 75 and Over and Their Caregivers
Acronym: CUIDAMOS+75
Status: Completed | Type: Observational
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital del Mar Research Institute (IMIM) (Other); Fundación para la Investigación e Innovación Biosanitaria de la Comunidad de Madrid (Unknown)
Responsible Party: Principal Investigator, Milagros Rico Blazquez, Principal researcher, Gerencia de Atención Primaria, Madrid
Other Study IDs: 20210009; PI21_00190 (Other Grant/Funding Number: Instituto de Salud Carlos III and ERDF); PI21_00648 (Other Grant/Funding Number: Instituto de Salud Carlos III and ERDF); PI21_CIII00015 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2022-02-08; First posted 2022-02-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-09

CONDITIONS: Aging; SARS-CoV-2 Infection; Caregivers; Frailty; Burden, Caregiver
Keywords: Aging; SARS-CoV-2 infection; Caregivers; Primary Health Care; Nursing process; Standardized Nursing Terminology; Health Services Research; Cohort Studies; Qualitative Research; Real world data; quality of life
MeSH Terms: conditions — COVID-19; Frailty; Caregiver Burden

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Infection: Confirmed SARS-CoV-2 infection diagnosed after 11 May 2020 and registered in electronic health records.
  (positive confirmatory test on nucleic acid amplification (rRT-PCR) or having had symptoms for <5 days is positive on a PRAg test)
  Interventions: Other: Exposure SARS-CoV-2 Infection
- NO SARS-CoV-2 Infection: No confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020.

INTERVENTIONS:
Other: Exposure SARS-CoV-2 Infection — The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020.
  Positive confirmatory test on nucleic acid amplification (rRT-PCR) or having had symptoms for <5 days is positive on a PRAg test.
  Groups: SARS-CoV-2 Infection

SUMMARY:
The measures to control the transmissibility of the Covid-19 pandemic have changed the daily routines of the population, increasing sedentary lifestyles, decreasing outdoor physical activity and limiting contact with neighbors, family and friends. This could be having negative consequences for the health of vulnerable people.

The investigators want to know how this situation has affected the health of people aged 75 years or older and their caregivers and how the circumstances experienced may mark new care needs.

To this end, will be analyzed clinical data, follow up people who have become ill with COVID-19 and those who have not, and interview groups of caregivers and patients to hear about the personal impact of the pandemic on them.

This will allow us to explore what changes are needed in health care to achieve an improvement in the health and quality of life of this population.

CUIDAMOS+75 seeks the commitment of the population and of the different people in charge of the health services from the very beginning.

DETAILED DESCRIPTION:
Objective:

To explore the impact of the pandemic SARS-CoV-2 on the state of health of people aged ≥75 years.

Design:

Mixed-methods study. 1) Multipurpose, ambispective, longitudinal population-based cohort study with real world data and 6 years of follow-up; 2) Prospective observational cohort study with 18 months of follow-up; 3) Qualitative study with a critical-social approach. Scope:

Primary care in 11 Autonomous Regions.

Population:

People aged ≥75 years, attending healthcare centres in the study area.

Sample:

The population cohort will include the total population that meets the criteria, out of the estimated 1619620. The prospective cohort size is 1035, recruited on a probabilistic basis by clinical nurses. In the social critical approach the selection will be intentional and will progress towards theoretical sampling according to the emerging findings.

V. outcome:

Population-based cohort: nursing diagnostic and interventions and use of services; mortality, quality of life (EQ-5D) and functional capacity (Barthel) for cohort follow-up.

V. exposure:

SARS-CoV-2 infection.

Sources:

Clinical history, clinical interview, semi-structured interviews and focus groups.

Analysis:

Population cohort: to explore the evolution of diagnostic and interventions, a time series analysis will be carried out. Cohort study: Kaplan-Meier survival curves for mortality, functional change and quality of life. Cox proportional hazards models will be used to study the impact of infection on the three variables at 6, 12 and 18 months, adjusted for socio-demographic and clinical variables. Qualitative study: thematic, semiotic and discursive positions analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one entry in the electronic medical record during 2018 (Sub-study 1).
* Have at least one entry in the clinical history during the last 6 months of 2019 (Sub-study 2).
* Give informed consent (Sub-study 2 & 3).
* Family caregivers of dependent persons included in the population cohort (Sub-study 3).

Exclusion Criteria:

* Not belonging to National Health System centres in the territorial demarcations participating in the study (Sub-study 1).
* Not belonging to the quotas of the 105 participating nurses (Sub-study 2 & 3).
* Carers who have been caring for less than 6 months at the start of the pandemic, with sensory or cognitive deficits (Sub-study 3).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Persons ≥75 years of age registered at the health centres in the study area. A total population of 1,619,620 users is estimated.
Sampling Method: Probability Sample
Enrollment: 1035 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Changes caused by the SARS-CoV-2 pandemic in the use of health services in a population-based cohort of non-institutionalised people aged 75 years and older. | up to 1 year
  By analysing real-life data from electronic clinical records.

SECONDARY OUTCOMES:
Changes from baseline prevalence of care needs of non-institutionalised people aged 75 and over in the context of the SARS-CoV-2 pandemic. | at the basal time.
  Sub-study 1: Longitudinal study of a population-based, multipurpose, ambispective cohort. Variables on nursing interventions will be collected through the primary care electronic medical record.
Changes from baseline prevalence of care needs of non-institutionalised people aged 75 and over in the context of the SARS-CoV-2 pandemic. | 6 years follow-up.
  Sub-study 1: Longitudinal study of a population-based, multipurpose, ambispective cohort. Variables on nursing interventions will be collected through the primary care electronic medical record.
Number of participants with changes caused by the SARS-CoV-2 pandemic in the functional capacity of non-institutionalised people aged 75 and over. | 18 months follow-up
  Sub-study 2: Prospective observational cohort study with a follow-up of 18 months. The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020. Data on change in functioning will be collected using the Barthel scale.
Number of participants with changes caused by the SARS-CoV-2 pandemic in the quality of life of non-institutionalised people aged 75 and over. | 18 months follow-up
  Sub-study 2: Prospective observational cohort study with a follow-up of 18 months. The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020. Data on change quality of life will be collected using the EQ-5D.
Number of participants with changes caused by the SARS-CoV-2 pandemic in the cognitive capacity of non-institutionalised people aged 75 years and over. | 18 months follow-up
  Sub-study 2: Prospective observational cohort study with a follow-up of 18 months. The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020. Data on change cognitive capacity will be collected using the Mini Mental Status Examination.
Number of participants with changes caused by the SARS-CoV-2 pandemic in the mental health of non-institutionalised people aged 75 and over. | 18 months follow-up
  Sub-study 2: Prospective observational cohort study with a follow-up of 18 months. The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020. Data on mental health capacity will be collected using the Hamilton Scale.
Incidence of mortality caused by the SARS-CoV-2 pandemic among non-institutionalised persons aged 75 years and over. | 18 months follow-up
  Sub-study 2: Prospective observational cohort study with a follow-up of 18 months. The exposure variable is confirmed SARS-CoV-2 infection with diagnosis after 11 May 2020. Mortality data shall be studied through medical records.
Understand and interpret the social, political and economic dimensions linked to the use of health services by people aged 75 and over and family caregivers during the pandemic and think about possible coping strategies. | zero time, baseline.
  Sub-study 3:Qualitative study with a social critical approach through semi-structured interviews for ≥75 years and focus groups for caregivers. A thematic analysis will be carried out, which will be complemented at the textual level by a semiotic analysis of discursive positions. In accordance with the critical character, discourse will be analysed as a reflection of ideological positions of inequality and domination.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rico-Blázquez, Master, Study Director — Gerencia Asistencial de Atención Primaria de Madrid
Locations (2):
- Spain (2):
  - Milagros Rico-Blazquez, Madrid, Madrid
  - Milagros Rico-Blázquez, Madrid, Madrid

REFERENCES:
- [Background] Alfano V, Ercolano S. The Efficacy of Lockdown Against COVID-19: A Cross-Country Panel Analysis. Appl Health Econ Health Policy. 2020 Aug;18(4):509-517. doi: 10.1007/s40258-020-00596-3. PMID 32495067
- [Background] Borges-Machado F, Barros D, Ribeiro O, Carvalho J. The Effects of COVID-19 Home Confinement in Dementia Care: Physical and Cognitive Decline, Severe Neuropsychiatric Symptoms and Increased Caregiving Burden. Am J Alzheimers Dis Other Demen. 2020 Jan-Dec;35:1533317520976720. doi: 10.1177/1533317520976720. PMID 33295781
- [Background] Brown EE, Kumar S, Rajji TK, Pollock BG, Mulsant BH. Anticipating and Mitigating the Impact of the COVID-19 Pandemic on Alzheimer's Disease and Related Dementias. Am J Geriatr Psychiatry. 2020 Jul;28(7):712-721. doi: 10.1016/j.jagp.2020.04.010. Epub 2020 Apr 18. PMID 32331845
- [Background] Cohen G, Russo MJ, Campos JA, Allegri RF. Living with dementia: increased level of caregiver stress in times of COVID-19. Int Psychogeriatr. 2020 Nov;32(11):1377-1381. doi: 10.1017/S1041610220001593. Epub 2020 Jul 30. PMID 32729446
- [Background] Company-Sancho MC, Estupinan-Ramirez M, Sanchez-Janariz H, Tristancho-Ajamil R. The connection between nursing diagnosis and the use of healthcare resources. Enferm Clin. 2017 Jul-Aug;27(4):214-221. doi: 10.1016/j.enfcli.2017.04.002. Epub 2017 May 10. English, Spanish. PMID 28501464
- [Background] Dubey S, Biswas P, Ghosh R, Chatterjee S, Dubey MJ, Chatterjee S, Lahiri D, Lavie CJ. Psychosocial impact of COVID-19. Diabetes Metab Syndr. 2020 Sep-Oct;14(5):779-788. doi: 10.1016/j.dsx.2020.05.035. Epub 2020 May 27. PMID 32526627
- [Background] Freijomil-Vazquez C, Gastaldo D, Coronado C, Movilla-Fernandez MJ. When risk becomes illness: The personal and social consequences of cervical intraepithelial neoplasia medical surveillance. PLoS One. 2019 Dec 16;14(12):e0226261. doi: 10.1371/journal.pone.0226261. eCollection 2019. PMID 31841543
- [Background] Holt-Lunstad J, Smith TB, Baker M, Harris T, Stephenson D. Loneliness and social isolation as risk factors for mortality: a meta-analytic review. Perspect Psychol Sci. 2015 Mar;10(2):227-37. doi: 10.1177/1745691614568352. PMID 25910392
- [Background] Johnson VR, Jacobson KL, Gazmararian JA, Blake SC. Does social support help limited-literacy patients with medication adherence? A mixed methods study of patients in the Pharmacy Intervention for Limited Literacy (PILL) study. Patient Educ Couns. 2010 Apr;79(1):14-24. doi: 10.1016/j.pec.2009.07.002. Epub 2009 Aug 3. PMID 19647967
- [Background] Lam K, Lu AD, Shi Y, Covinsky KE. Assessing Telemedicine Unreadiness Among Older Adults in the United States During the COVID-19 Pandemic. JAMA Intern Med. 2020 Oct 1;180(10):1389-1391. doi: 10.1001/jamainternmed.2020.2671. PMID 32744593
- [Background] Lamont RA, Nelis SM, Quinn C, Clare L. Social Support and Attitudes to Aging in Later Life. Int J Aging Hum Dev. 2017 Jan;84(2):109-125. doi: 10.1177/0091415016668351. Epub 2016 Sep 20. PMID 27655953
- [Background] Mann DM, Chen J, Chunara R, Testa PA, Nov O. COVID-19 transforms health care through telemedicine: Evidence from the field. J Am Med Inform Assoc. 2020 Jul 1;27(7):1132-1135. doi: 10.1093/jamia/ocaa072. PMID 32324855
- [Background] Mowbray H. In Beijing, coronavirus 2019-nCoV has created a siege mentality. BMJ. 2020 Feb 7;368:m516. doi: 10.1136/bmj.m516. No abstract available. PMID 32033967
- [Background] Perez-Rodrigo C, Gianzo Citores M, Hervas Barbara G, Ruiz-Litago F, Casis Saenz L, Arija V, Lopez-Sobaler AM, Martinez de Victoria E, Ortega RM, Partearroyo T, Quiles-Izquierdo J, Ribas-Barba L, Rodriguez-Martin A, Salvador Castell G, Tur JA, Varela-Moreiras G, Serra-Majem L, Aranceta-Bartrina J. Patterns of Change in Dietary Habits and Physical Activity during Lockdown in Spain Due to the COVID-19 Pandemic. Nutrients. 2021 Jan 21;13(2):300. doi: 10.3390/nu13020300. PMID 33494314
- [Background] Roschel H, Artioli GG, Gualano B. Risk of Increased Physical Inactivity During COVID-19 Outbreak in Older People: A Call for Actions. J Am Geriatr Soc. 2020 Jun;68(6):1126-1128. doi: 10.1111/jgs.16550. Epub 2020 May 14. No abstract available. PMID 32392620
- [Background] Saltzman LY, Pat-Horenczyk R, Lombe M, Weltman A, Ziv Y, McNamara T, Takeuchi D, Brom D. Post-combat adaptation: improving social support and reaching constructive growth. Anxiety Stress Coping. 2018 Jul;31(4):418-430. doi: 10.1080/10615806.2018.1454740. Epub 2018 Apr 12. PMID 29649912
- [Background] Saltzman LY, Hansel TC, Bordnick PS. Loneliness, isolation, and social support factors in post-COVID-19 mental health. Psychol Trauma. 2020 Aug;12(S1):S55-S57. doi: 10.1037/tra0000703. Epub 2020 Jun 18. PMID 32551762
- [Derived] Rico-Blazquez M, Esteban-Sepulveda S, Sanchez-Ruano R, Aritztegui-Echenique AM, Artigues-Barbera EM, Brito-Brito PR, Casado-Ramirez E, Cidoncha-Moreno MA, Fabregat-Julve MI, Feria-Raposo I, Hernandez-Pascual M, Lozano-Hernandez C, Moreno-Casbas MT, Otones-Reyes P, Palmar-Santos AM, Pedraz-Marcos A, Romero-Rodriguez EM, Sole-Agusti MC, Taltavull-Aparicio JM, Vidal-Thomas MC, Gonzalez-Chorda VM; Cuidamos+75 Group. Impact of the COVID-19 pandemic on the self-care and health condition of the older adults. CUIDAMOS+75. A mixed methods study protocol. Front Public Health. 2024 Jun 17;12:1389641. doi: 10.3389/fpubh.2024.1389641. eCollection 2024. PMID 38952731